CLINICAL TRIAL: NCT05465538
Title: Effect of Cannabis Use on Synaptic Density in Older Adults
Brief Title: SV2A in Older Adults
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Principal Investigator, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000032183
Record Dates: First submitted 2022-07-16; First posted 2022-07-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Cannabis Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabis using older adults (Other): Subjects undergo a single PET scan using [11C]UCB-J
  Interventions: Drug: [11C]UCB-J PET
- Healthy controls (Other): Subjects undergo a single PET scan using [11C]UCB-J
  Interventions: Drug: [11C]UCB-J PET

INTERVENTIONS:
Drug: [11C]UCB-J PET — Single PET scan using the radioligand [11C]UCB-J

SUMMARY:
The aim of the study is to examine the effect of cannabis use on brain synaptic density among older adults using [11C]UCB-J PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Male or female, aged ≥50 years
* No history of significant medical or neurological disease
* BMI ≤ 50
* If woman of childbearing potential, must agree to use an acceptable method of birth control, as determined by the principal investigator, for the duration of the study and up to one month after completion of PET scans

Exclusion Criteria:

* Women with a positive pregnancy test or women who are lactating
* Have had exposure to ionizing radiation that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits;
* History of a bleeding disorder or are currently taking anticoagulants
* Subjects who have donated blood within 8 weeks of the present study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hippocampal synaptic density | 1 month
  Measure of synaptic density in the hippocampus

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MBBS, MD, Principal Investigator — Yale University
Locations (1):
- Conneticut Mental Health Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No